CLINICAL TRIAL: NCT06144424
Title: Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of EP262 in Subjects With Atopic Dermatitis (EASE)
Brief Title: Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of EP262 in Subjects With Atopic Dermatitis
Acronym: EASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Escient Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-262-202
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EP262 150 mg (Experimental)
  Interventions: Drug: Oral EP262
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral EP262 — Once daily
  Arms: EP262 150 mg
Drug: Placebo — Once Daily
  Arms: Placebo

SUMMARY:
This Phase 2a trial will evaluate the effects of EP262 in subjects with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of active atopic dermatitis for at least 1 year
* BSA of 3% to 20% and a vIGA-AD score of ≥3

Exclusion Criteria:

* Other active skin diseases associated with chronic pruritus
* Clinically infected atopic dermatitis that requires antibiotic therapy
* Use of specific treatments for atopic dermatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Allervie Clinical Research, Birmingham, Alabama
  - RM Medical Research, Inc., Miami Lakes, Florida
  - Indiana Clinical Trials Center, Plainfield, Indiana
  - Lawrence J. Green, MD LLC, Rockville, Maryland
  - Revival Research Institute, LLC, Troy, Michigan
  - Optima Research Boardman, Boardman, Ohio
  - J&S Studies, Inc., College Station, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Dermatology Specialists of Spokane, Spokane, Washington
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in the United States and Canada.
Groups:
- 150 mg EP262 QD: Participants received oral EP262 150 milligrams (mg) QD during the 6-week Double-blind Treatment Period. After administration of the last dose, participants entered a 4-week Follow-up Period.
- Placebo QD: Participants received matching oral placebo once daily (QD) during the 6-week Double-blind Treatment Period. After administration of the last dose, participants entered a 4-week Follow-up Period.
Period: Overall Study
Arm/Group | 150 mg EP262 QD | Placebo QD
Started | 21 | 11
Completed | 18 | 11
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Incarceration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg EP262 QD | Placebo QD | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (16.54) | 41.7 (11.30) | 40.3 (14.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 18 | 11 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black or African American | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. A TEAE is defined as an adverse event (AE) with an onset after the first dose of study drug or an existing event that worsened after the first dose during the study.
Time Frame: up to Week 10
Population: Safety Analysis Set: all participants who were randomized and took at least 1 dose of randomized study drug. Safety analyses were based upon treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg EP262 QD | Placebo QD
Number analyzed (Participants) | 21 | 11
Participants | 4 | 7

2. Primary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. A TEAE is defined as an adverse event (AE) with an onset after the first dose of study drug or an existing event that worsened after the first dose during the study. AEs were graded for severity using the the Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v.5). CTCAE grades were scored as: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe or medically significant; Grade 4 = life threatening; Grade 5 = death related to the AE.
Time Frame: up to Week 10
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg EP262 QD | Placebo QD
Number analyzed (Participants) | 21 | 11
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Vital Signs
Description: Clinical meaningfulness was determined by the investigator.
Time Frame: up to Week 10
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg EP262 QD | Placebo QD
Number analyzed (Participants) | 21 | 11
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Electrocardiograms (ECGs )
Description: Clinical meaningfulness was determined by the investigator.
Time Frame: up to Week 10
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg EP262 QD | Placebo QD
Number analyzed (Participants) | 18 | 11
Participants | 1 | 1

5. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Clinical Hematology, Chemistry, or Coagulation Parameters
Description: Clinical meaningfulness was determined by the investigator.
Time Frame: up to Week 10
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg EP262 QD | Placebo QD
Number analyzed (Participants) | 21 | 11
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With a Change From Baseline to Week 6 in Gene Expression Signature and Skin Histology (Epidermal Thickness, Immune Cell Infiltration, Markers of Epidermal Proliferation) as Assessed From Biopsies of Lesional Skin
Description: Biopsies were taken from lesional and nonlesional skin, and differential gene expression was analyzed by comparing lesional samples at baseline and Week 6 to nonlesional reference samples at baseline. Genes were classified as differentially expressed if they met 2 criteria: an absolute log2 fold change greater than 1.5 and an adjusted p-value less than 0.05 using Wilcoxon signed rank test or paired Students t-test and Bonferroni correction.
Time Frame: Baseline; Week 6
Population: Full Analysis Set: all participant who were randomized and took at least 1 dose of randomized study drug. Participants were analyzed according to randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg EP262 QD | Placebo QD
Number analyzed (Participants) | 21 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to Week 10
Description: Analysis was conducted in the Safety Analysis Set, comprised of all participants who were randomized and took at least 1 dose of randomized study drug. Safety analyses were based upon treatment actually received.
Arm/Group | Placebo QD | 150 mg EP262 QD
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/21
Other Adverse Events (participants affected / at risk) | 7/11 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QD (N=11) | 150 mg EP262 QD (N=21)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral rash (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT06144424/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT06144424/SAP_001.pdf